CLINICAL TRIAL: NCT03675542
Title: A Phase 1b, Open-label, Single-arm, Dose-selection, Proof-of-concept Study to Assess the Safety and Efficacy of a Novel HSP90 Inhibitor (CUDC-305) in the Treatment of Moderate to Severe Plaque Psoriasis
Brief Title: The Safety and Efficacy of a Novel HSP90 Inhibitor (CUDC-305) in the Treatment of Moderate to Severe Psoriasis.
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Aarhus University Hospital (Other)
Responsible Party: Principal Investigator, Anne Bregnhøj, Principal Investigator, Aarhus University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CUDC305
Record Dates: First submitted 2018-09-17; First posted 2018-09-18 (Actual); Last update posted 2019-07-11 (Actual); Status verified 2019-07

CONDITIONS: Psoriasis Vulgaris
MeSH Terms: interventions — CUDC 305

STUDY DESIGN:
Intervention Model Description: open-label, singlecenter, single-arm, dose-selection, proof of-concept study
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Study medication (Experimental): HSP90 inhibitor (CUDC-305)
  Interventions: Drug: CUDC-305

INTERVENTIONS:
Drug: CUDC-305 — Dose-selection treatment with HSP90 inhibitor (CUDU-305)

SUMMARY:
This is a 12-week treatment, singlecenter, open-label, single-arm, dose-selection, proof of concept study to determine a dosage of HSP 90 inhibitor (CUDC-305) that is tolerable and demonstrates preliminary efficacy for use in future efficacy Phase 2 trials. Male or female subjects aged 18 years or older with moderate to severe plaque psoriasis will be included in this study.

Objectives are to determine the efficacy, safety and tolerability of CUDC-305 in patients with moderate to severe psoriasis.

ELIGIBILITY:
Inclusion Criteria:

1. Men or women aged 18 years or older at the time of consent.
2. Subject has a history of plaque psoriasis for at least 6 months prior to the screening visit.
3. Subject has stable psoriasis conditions for at least 3 months before screening, according to subject.
4. Subject has plaque psoriasis covering ≥3% of his total BSA at baseline (Day 0).
5. Subject has a PASI score of ≥6 at baseline (Day 0).
6. Subject has a PGA score of ≥3 at baseline (Day 0).
7. Subject has a body mass index (BMI) ≤40 kg/m2.
8. Subject is a candidate for phototherapy or systemic treatement of psoriasis (either naïve or has a history of previous treatment).
9. Subjects (women and men) involved in any sexual intercourse that could lead to pregnancy must agree to use an effective contraceptive method from at least 4 weeks before baseline (Day 0) until at least 4 weeks after the last study product administration for the duration of the study. Effective contraceptive methods are: systemic hormonal contraceptives (oral contraceptive, patch, vaginal ring, injectables, or implants), intrauterine devices, vasectomy, or barrier methods of contraception in conjunction with spermicide. Hormonal contraceptives must be on a stable dose for at least 4 weeks before baseline (Day 0).

   Note: Women of nonchildbearing potential are as follows:
   * Women who have had surgical sterilization (hysterectomy, bilateral oophorectomy, bilateral salpingectomy, or bilateral tubal ligation)
   * Women ≥60 years of age
   * Women >40 and <60 years of age who have had a cessation of menses for at least 12 months and a follicle-stimulating hormone (FSH) test confirming nonchildbearing potential (FSH ≥40 mIU/mL) or cessation of menses for at least 24 months without FSH levels confirmed
10. Women of childbearing potential must have a negative serum pregnancy test at screening and negative urine pregnancy test at baseline (Day 0).
11. Subject must have negative tuberculosis (TB) infection tests. Subject will be evaluated for latent TB infection with a purified protein derivative (PPD) test, T-spot test or a Quantiferon Gold test, and with a chest x-ray, if one has not been performed in the last 6 months. Subject who demonstrates evidence of latent TB infection (either PPD greater than or equal to 5 mm of induration or positive Quantiferon Gold or T-spot test, irrespective of Bacillus Calmette-Guérin (BCG) vaccination status and negative chest x ray findings for active TB, or suspicious chest x-ray findings) will not be allowed to participate in the study.
12. Subject must be willing to participate and must be capable of giving informed consent, and the consent must be obtained prior to any study-related procedures.

Exclusion Criteria:

1. Female subject who is breastfeeding, pregnant, or who is planning a pregnancy during the study.
2. Subject has evidence of erythrodermic, pustular, predominantly guttate psoriasis, or drug induced psoriasis.
3. Subject has a history of skin disease or presence of skin condition that, in the opinion of the investigator, would interfere with the study assessments.
4. Subject is known to have immune deficiency or is immunocompromised.
5. Subject has a history of cancer or lymphoproliferative disease within 5 years prior to baseline (Day 0). Subjects with successfully treated non-metastatic cutaneous squamous cell or basal cell carcinoma and/or localized carcinoma in situ of the cervix are not to be excluded.
6. Subject has had a major surgery within 8 weeks prior to baseline (Day 0) or has a surgery planned during the study.
7. Subject has any clinically significant medical condition or physical/laboratory/ECG/vital signs abnormality that would, in the opinion of the investigator, put the subject at undue risk or interfere with interpretation of study results.
8. Subject has alanine aminotransferase (ALT) or aspartate aminotransferase (AST) values ≥ 2 times the upper limit of normal (ULN) at screening.
9. Subject has absolute neutrophil count ≤1,5 X 109/L or platelet count ≤100 X 109/L at screening.
10. Subject has history of clinically significant anemia or hemoglobin (Hgb) value ≤ 10 g/dL at screening.
11. Subject has a creatinine clearance ≤ 60 ml/min at screening (calculated with Cockcroft-Gault formula)
12. Subject with positive results for hepatitis B surface antigens (HBsAg), anti-hepatitis B core antibodies (anti-HBc), hepatitis C virus (HCV), or human immunodeficiency virus (HIV).
13. Subject has a known or suspected allergy to CUDC-305 or any component of the investigational product.
14. Subject has a history of clinically significant drug or alcohol abuse in the last year prior to baseline visit (Day 0).
15. Subject is currently receiving an investigational product or device or has received one within 4 weeks prior to baseline visit (Day 0).
16. Subject has used biologics medication 12 weeks prior to baseline visit (Day 0), or 5 half lives (whichever is longer).
17. Subject has used any systemic treatment for psoriasis (including corticosteroids, oral retinoids, immunosuppressive medication, methotrexate, cyclosporine, or apremilast) within 4 weeks prior to baseline visit (Day 0).
18. Subject has used any topical medication to treat psoriasis (including corticosteroids; retinoids; vitamin D analogues, such as calcipotriol; or tar) within 2 weeks prior to baseline visit (Day 0).
19. Subject had any UVB phototherapy (including tanning beds) or excimer laser within 2 weeks prior to baseline visit (Day 0).
20. Subject had PUVA treatment within 4 weeks prior to baseline visit (Day 0).
21. Subject has received a live attenuated vaccine within 4 weeks prior to baseline visit (Day 0) or plan to receive a live attenuated vaccine during the study and up to 1 month after the last study drug administration.Subject had excessive sun exposure within 2 weeks prior to baseline visit (Day 0), or is planning a trip to a sunny climate, or is not willing to minimize natural and artificial sunlight exposure during the study. Use of sunscreen products and protective apparel are recommended for other circumstances when exposure cannot be avoided. Sunscreen must not be applied on the clinic visit days before the visit.
22. Subject has a history of an allergic reaction or significant sensitivity to lidocaine or other local anesthetics.
23. Subject has a history of hypertrophic scarring or keloid formation in scars or suture sites.
24. Subject is taking anticoagulant medication, such as heparin, low molecular weight (LMW) heparin, warfarin, antiplatelets (nonsteroidal anti-inflammatory drugs [NSAIDs] and low-dose aspirin that is equal or lower than 81 mg will not be considered antiplatelets), or has a contraindication to skin biopsies.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2018-11-01 (Actual); Primary Completion 2019-11-01 (Estimated); Study Completion 2020-02-01 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in Psoriasis Area and Severity Index (PASI) score | Week 12
  Clinical severity score

SECONDARY OUTCOMES:
Incidence of treatment-emergent adverse events (TEAEs) | Week 12
  TEAEs

CONTACTS AND LOCATIONS:
Locations (1):
- Aarhus University Hospital, Aarhus, Denmark

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol (2018-06-22): https://cdn.clinicaltrials.gov/large-docs/42/NCT03675542/Prot_000.pdf